CLINICAL TRIAL: NCT03174028
Title: Laparoscopically Assisted Anorectal Pull-through Versus Posterior Sagittal Anorectoplasty for High and Intermediate Anorectal Malformations : A Comparative Study
Brief Title: Laparoscopically Assisted Anorectal Pull-through Versus Posterior Sagittal Anorectoplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Gamal Abdelmalek, principle investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: lAR
Record Dates: First submitted 2017-05-30; First posted 2017-06-02 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Anorectal Malformation
MeSH Terms: conditions — Anorectal Malformations

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic group (Active Comparator): laparoscopic pull-through
  Interventions: Device: laparoscopic pull-through
- posterior sagittal group (Sham Comparator): posterior sagittal anorectoplasty
  Interventions: Device: laparoscopic pull-through

INTERVENTIONS:
Device: laparoscopic pull-through — laparoscopic pull-through

SUMMARY:
Anorectal malformations are congenital malformations, in which the terminal part of the hindgut is abnormally placed and lies outside (partially or completely) the sphincter mechanism.

DETAILED DESCRIPTION:
The incidence of anorectal malformation ~1 in 5,000 More common in Down's syndrome and Cat-eye syndrome. Male >female (60:40).It is classified into many types according to the degree of descent of the rectal pouch in the pelvis, the fistula between the rectum and the urinary system in males and genital system in females. The most common type in males is high anorectal malformation with rectourethral fistula

There are many historical operations for the management of the high type, but the most popular operation now is the posterior sagittal anorectoplasty which was published for the first time in 1982. Children undergoing posterior sagittal anorectoplasty may have lifelong bowel management problems of constipation, incontinence, and encopresis.

After the introduction of laparoscopy in pediatric surgery, many surgeons hope that the use of laparoscopy instead of posterior sagittal anorectoplasty may reduce the complications of the complications of the big incision and disturbance of sphincter mechanism which occur in posterior sagittal anorectoplasty operation. In addition to its role in diagnosis in complex anomalies like cloaca which is well established now. So the question is to what extent can the laparoscopy replace usual surgery for anorectal malformation.

ELIGIBILITY:
Inclusion Criteria:

-all male and female childs aged from 6 months to the age of 3 years, in assiut university hospital, who have been diagnosed to have high anorectal malformation since birth and for whom colostomy was done

Exclusion Criteria:

* all cases with low anomalies will be excluded.
* Female child with vestibular anus
* case with short distal pouch

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
stool continence | 3 months
  questionaire about the degree of stool continence

IPD SHARING:
Plan to Share IPD: No